CLINICAL TRIAL: NCT04987021
Title: An Actual Use, Prospective, Adaptive Design, Single Centre, Non-randomised, Open-label Study, Assessing Usability of Remote Assist When Used to Program Cochlear Implant Recipients
Brief Title: An Actual Use, Open-label Study Assessing Usability of Remote Assist to Program Cochlear Implant Recipients
Acronym: RAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CLTD5809
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-07

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral
Keywords: Cochlear Implant; Remote Programming; Tele-audiology; Tele-medicine
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nucleus Smart App with Remote Assist Custom Sound Pro 6.3 (Experimental): Remote Assist Custom Sound Pro 6.3 to enable clinicians to use the App to remotely to program the recipients sound processors.
  Interventions: Device: Cochlear Implant (CI)-CI500 series, CI600 series or Freedom series cochlear implants

INTERVENTIONS:
Device: Cochlear Implant (CI)-CI500 series, CI600 series or Freedom series cochlear implants — The Remote Assist (RA) System is intended to support clinicians to conduct a remote programming session with their CI recipients.

SUMMARY:
Clinical management of cochlear implant (CI) recipients involve programming, counselling, performance evaluation and habilitation. This requires the recipients to travel to the clinic for follow up appointments which can pose significant challenges for recipients, particularly those who live far away from the clinic. Remote Assist (RA) is a new solution that allows the clinician to make MAP and sound processor adjustments via the recipient's Nucleus Smart app (NSA) installed on their smart phone. With RA the clinician can also perform counselling using a video call directly via the NSA. As RA uses no specialized hardware and software that needs to be sent and retrieved back from the recipient, it has the potential to further improve the remote programming experience and convenience for both the recipient and the clinician.

DETAILED DESCRIPTION:
Clinical management of cochlear implant (CI) recipients involve programming, counselling, performance evaluation and habilitation. The standard practice for this management involves frequent clinical visits in the first year after implantation and annual visits for the rest of the recipient's life. The need to travel to the clinic for follow up appointments can pose significant challenges for recipients, particularly those who live far away from the clinic. There have been reports of recipients being lost to follow up due to the difficulties in travelling to the clinic. The inconvenience of scheduling a session and travelling to the clinic might deter recipients from seeking help for some seemingly small / less troubling issues and increase their tendency to somehow bear and live with the issues. Sometimes clinicians schedule follow-up sessions with the primary purpose of following-up on progress with strategies provided earlier to overcome real world problems. Such follow-up on progress can easily be completed via a video call as well. Remote programming is one telehealth solution known to be successful in addressing the challenges of travelling to the clinic for appointments. During the Covid-19 pandemic there was a demonstrated increase in the uptake of remote programming when traveling to the clinic posed a health and safety risk. Current methods of remote programming of CI requires the use of special computer and programming hardware as well as proprietary programming software to be installed on a personal computer (PC) at the remote location. Although remote programming potentially reduces the travel burden for some recipients, it involves substantial administrative effort and cost by clinics to prepare, send, retrieve back, and clean remote programming hardware and software. This also reduces the frequency with which remote programming appointments can be scheduled due to time delays in sending and retrieving equipment. Remote Assist (RA) is a new solution that allows the clinician to make MAP and sound processor adjustments via the recipient's Nucleus Smart app (NSA) installed on their smart phone. With RA the clinician can also perform counselling using a video call directly via the NSA. As RA uses no specialized hardware and software that needs to be sent and retrieved back from the recipient, it has the potential to further improve the remote programming experience and convenience for both the recipient and the clinician.

The current study aims to assess recipients ease and experience with using Remote Assist to receive remote programming of their CI.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years).
2. Implanted with the below cochlear implants in one or both ears. CI500 series (CI512, CI513, CI522, CI532,), CI600 series (CI612, CI622, CI632), Freedom series (CI24RE (ST), CI24RE (CA), CI24RE (CS), CI422).
3. At least 3 months experience with the cochlear implant.
4. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
2. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
3. Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
4. Currently participating or participated in another interventional clinical study/trial in the past 30 days, or if less than 30 days the prior investigation was Cochlear sponsored and determined by the investigator to not impact clinical findings of this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cochlear Sydney In-house lab, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nucleus Smart App With Remote Assist Custom Sound Pro 6.3
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nucleus Smart App With Remote Assist Custom Sound Pro 6.3
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 63 [44 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 15
Age at test [Median (Full Range); unit: years] | 63 [44 to 90]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who While Using the Final Version of Remote Assist, Are Able to Complete the Primary Tasks (Score of 5 on the Usability Rating Scale)
Description: Usability rating scale: 1 = unable to complete; 2 = Completed after help using document; 3 = Completed after trying an incorrect option; 4 = Completed after some exploration; 5 = Complete at first attempt.
Time Frame: Immediately after the participants´ first use of the Nucleus Smart App with Remote Assist Custom Sound Pro 6.3, on average half an hour after participants have completed all tasks.
Measure: Count of Participants; unit: Participants
Arm/Group | Nucleus Smart App With Remote Assist Custom Sound Pro 6.3
Number analyzed (Participants) | 15
Participants | 13

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | Nucleus Smart App With Remote Assist Custom Sound Pro 6.3
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nucleus Smart App With Remote Assist Custom Sound Pro 6.3 (N=15)
Sound levels uncomfortably loud (Investigations) | 1 (1) — One participant experienced an adverse device effect (ADE) of sounds being uncomfortably loud when being programmed with RA. The Adverse event resolved when stimulation using the IMD was stopped

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT04987021/Prot_SAP_000.pdf